CLINICAL TRIAL: NCT04058002
Title: Project Arthritis Recovering Quality of Life Through Education 70+
Acronym: PARQVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marcia Uchoa Rezende, Full Professor in Orthopedics and Traumatology, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 04019418.7.0000.0068
Record Dates: First submitted 2019-06-26; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee; Quality of Life; Sarcopenia
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Multiprofessional treatment and Educational Program Associated (EPA+C+BCAA) with supplementation of creatine and BCAA.
  Interventions: Other: Multiprofessional treatment and Educational Program Associated (EPA+C+BCAA) with supplementation of creatine and BCAA.
- Control group (Active Comparator): Multiprofessional treatment and Educational Program Associated (EPA+C) with supplementation of creatine only.
  Interventions: Other: Multiprofessional treatment and Educational Program Associated (EPA+C) with supplementation of creatine only.

INTERVENTIONS:
Other: Multiprofessional treatment and Educational Program Associated (EPA+C+BCAA) with supplementation of creatine and BCAA. — 17 patients will participate in two days of lectures two-months apart on the subject of knee OA, but will also come to the hospital at months 1, 3 and 5 after the first class to consult about nutritional habits to be improved; at months 4 and 6 to participate in a group therapy session with the psychologists, 7 sessions with the physical therapy team followed by 7 sessions with the physical educators team (once a week/4 weeks and once every two weeks, three times). Patients will be supplemented with creatine 5 grams and maltodextrin 100g, 30 minutes before training. At breakfast they will also ingest 5 grams of BCAA (1,200 milligrams of leucine, 600 milligrams of isoleucine and 600 milligrams of valine per dose)
  Arms: Experimental
Other: Multiprofessional treatment and Educational Program Associated (EPA+C) with supplementation of creatine only. — 17 patients will participate in two days of lectures two-months apart on the subject of knee OA, but will also come to the hospital at months 1, 3 and 5 after the first class to consult about nutritional habits to be improved; at months 4 and 6 to participate in a group therapy session with the psychologists, 7 sessions with the physical therapy team followed by 7 sessions with the physical educators team (once a week/4 weeks and once every two weeks, three times). Patients will be supplemented with creatine 5 grams and maltodextrin 100g, 30 minutes before training. At breakfast they will also ingest 5 grams of placebo.
  Arms: Control group

SUMMARY:
Introduction: Quadriceps weakness was previously associated with functional impairment of osteoarthritis (OA). Evidence also suggests that muscle strength may prevent the progression of existing OA. It is estimated that the decline in muscle mass between 40 and 80 years is between 30% and 50%, with reported losses in functional capacity reaching 3% each year beyond the age of 60 years. Therefore, procedures capable of increasing the effects of exercise on muscle strength and function may be beneficial for elderly patients with knee OA. The results of our studies have shown that with each year of life the patient loses strength gain capacity. Objective: To evaluate if a multiprofessional educational program associated with BCAA and creatine supplementation improves the quality of life, function, pain and body composition of patients with OA and age greater than or equal to 70 years. METHODS: 34 patients with knee OA and age greater than or equal to 70 years will undergo an educational and physical training program lasting 20 weeks. Half of the patients will receive creatine (control) and the others will receive creatine and BCAA (study). Patients will be evaluated through functional tests (sit-up and 30-second tests and time up and go), standardized questionnaires (WOMAC and Lequesne), quality of life scales (Euroqol-EQ-5D-5L), pain (through VAS), body composition and bone density (through densitometry), and level of physical activity. All of the above parameters will be assessed at the beginning of the study and 6 and 12 months later. All project costs will be reported and a cost-effectiveness and cost-utility analysis will be performed. All project costs will be reported and a cost-effectiveness and cost-utility analysis will be performed.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common form of arthritis, affecting mainly women. Patients with OA present pain that usually worsens with weight support and improves with rest, as well as morning stiffness and after periods of inactivity.

Quadriceps weakness was previously associated with functional impairment of OA. Evidence also suggests that muscle strength may prevent the progression of existing OA. In fact, positive associations were found between increased quadriceps strength and self-efficacy of ambulation, reduction of pain and improvement of function, emphasizing the role of muscle strengthening in the treatment of knee OA.

It is estimated that the decline in muscle mass between 40 and 80 years is between 30% and 50%, with reported losses in functional capacity reaching 3% each year after the age of 60 years. Therefore, procedures capable of enhancing the effects of exercise on muscle strength and function may be beneficial for elderly patients with knee OA.

The results of our previous studies have shown that with each year of life the patient loses strength gain capacity.

Creatine is a natural amine endogenously synthesized by the liver, kidney and pancreas or obtained in the diet from red meat, seafood and dairy products. Creatine plays an important role in rapid energy supply, being stored mainly in the skeletal muscles (90%) as phosphocreatine, a high energy phosphate involved in the rapid resynthesis of adenosine triphosphate during muscle contraction. It has already been demonstrated that the combination of resistance training and creatine supplementation is superior to exercise alone in the elderly and has proved to be a useful tool in the elderly with knee OA.

Studies have demonstrated the need for a higher protein intake in the elderly with some studies showing greater protein synthesis and improved body composition parameters.

The investigators believe that an education and physical activity program, used in the previous work of the authors that presented improvement of WOMAC, that can be reproduced in any basic health care unit, along with supplementation with creatine and branched chain amino acids can lead to an improvement functional evaluation of elderly patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with OAJ with or without metabolic syndrome (ie at least two of: overweight / obese, hyperglycemia, dyslipidemia, hypertension)
* Age greater than or equal to 70 years.
* Classified as degrees I to III of Kelgreen and Lawrence (K-L), that is, any degree of gonarthritis without obliteration of joint space.
* Indication of clinical treatment of OA
* Patients without disabsorbing syndrome or inflammatory diseases of the gastrointestinal tract (GIT).
* Patients not undergoing gastroplasty or surgery that altered the transit of food in the TGI (Roux "Y", for example).
* Patients with creatinine clearance greater than 60 ml / min / 1.73m2
* Patients not submitted to previous arthroplasty in the lower limbs.
* Patients not submitted to infiltration in the knees up to 6 months before the study.
* Patients with no personal history of cognitive, psychiatric and / or neurological disorders, whose symptoms presented at the time of evaluation are related or significantly interfere with the functions of attention, memory, logical reasoning, comprehension, in order to impair the assimilation of the given guidelines.
* Ability to read, understand and respond to the questionnaires

Exclusion Criteria:

* Missing the schedules and not performing the tasks as performed by the professionals.
* Patients who develop allergy or intolerance to creatine, dextrose or BCAA during the study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-08-15 (Estimated); Primary Completion 2020-02-15 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Participants who improve function by performing the sit to stand 30 seconds test (STS30) | 6 months
  Compare supplementation with creatine and BCAA to supplementation with creatine only improves the functional results of patients in the sit to stand 30 seconds (STS30)

SECONDARY OUTCOMES:
Change of results in the sit to stand 30 seconds test | 12 months
  Perform sit to stand 30 seconds test, recording the number of stands a person can complete in 30 seconds, more fast better.
Change of results in the Time up and go test | 6 months and 12 months
  Perform time up and go test, The time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down, faster perform better.
Change of results in the Womac questionnaire | 6 months and 12 months
  Answer Womac Questionnaire - Ranges: minimum 0 (Better, no pain and limitation) / maximum 96 (Worst pain and limitation)
Change of results in the Lequesne questionnaire | 6 months and 12 months
  Answer Lequesne Questionnaire - Ranges: minimum 0 (Better, no limitation) / maximum 24 (Worst limitation)
Change of results in the Visual Analogue Scale | 6 months and 12 months
  Answer Visual Analogue Scale - Ranges: minimum 0 (Better, no pain) / maximum 100 (Worst pain)
Change of results in the EuroQol Scale | 6 months and 12 months
  Answer EuroQol Scale - Ranges: minimum 0 (Better) / maximum 2 (Worst)
Change fat percentage | 6 months and 12 months
  Calculate fat percentage
Change lean mass percentage | 6 months and 12 months
  Calculate lean mass

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme P Ocampos, MD, Principal Investigator — University of São Paulo General Hospital
Locations (1):
- Instituto de Ortopedia e Traumatologia do Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Recommendations for the medical management of osteoarthritis of the hip and knee: 2000 update. American College of Rheumatology Subcommittee on Osteoarthritis Guidelines. Arthritis Rheum. 2000 Sep;43(9):1905-15. doi: 10.1002/1529-0131(200009)43:93.0.CO;2-P. No abstract available. PMID 11014340
- [Background] Slemenda C, Brandt KD, Heilman DK, Mazzuca S, Braunstein EM, Katz BP, Wolinsky FD. Quadriceps weakness and osteoarthritis of the knee. Ann Intern Med. 1997 Jul 15;127(2):97-104. doi: 10.7326/0003-4819-127-2-199707150-00001. PMID 9230035
- [Background] Lange AK, Vanwanseele B, Fiatarone Singh MA. Strength training for treatment of osteoarthritis of the knee: a systematic review. Arthritis Rheum. 2008 Oct 15;59(10):1488-94. doi: 10.1002/art.24118. PMID 18821647
- [Background] Altman RD. Early management of osteoarthritis. Am J Manag Care. 2010 Mar;16 Suppl Management:S41-7. PMID 20297876
- [Background] Patel HP, Syddall HE, Jameson K, Robinson S, Denison H, Roberts HC, Edwards M, Dennison E, Cooper C, Aihie Sayer A. Prevalence of sarcopenia in community-dwelling older people in the UK using the European Working Group on Sarcopenia in Older People (EWGSOP) definition: findings from the Hertfordshire Cohort Study (HCS). Age Ageing. 2013 May;42(3):378-84. doi: 10.1093/ageing/afs197. Epub 2013 Feb 5. PMID 23384705
- [Background] Reaes FM, Ivo MMAA, Scarcella DDS, Almeida LC, Suzuki RM, Rezende MU. EFFECT OF THE P.A.R.Q.V.E ON RHIZARTHRITIS. Acta Ortop Bras. 2018 Jan-Feb;26(1):41-47. doi: 10.1590/1413-785220182601184420. PMID 29977144
- [Background] Wyss M, Kaddurah-Daouk R. Creatine and creatinine metabolism. Physiol Rev. 2000 Jul;80(3):1107-213. doi: 10.1152/physrev.2000.80.3.1107. PMID 10893433
- [Background] Gualano B, Macedo AR, Alves CR, Roschel H, Benatti FB, Takayama L, de Sa Pinto AL, Lima FR, Pereira RM. Creatine supplementation and resistance training in vulnerable older women: a randomized double-blind placebo-controlled clinical trial. Exp Gerontol. 2014 May;53:7-15. doi: 10.1016/j.exger.2014.02.003. Epub 2014 Feb 13. PMID 24530883
- [Background] Brose A, Parise G, Tarnopolsky MA. Creatine supplementation enhances isometric strength and body composition improvements following strength exercise training in older adults. J Gerontol A Biol Sci Med Sci. 2003 Jan;58(1):11-9. doi: 10.1093/gerona/58.1.b11. PMID 12560406
- [Background] Devries MC, Phillips SM. Creatine supplementation during resistance training in older adults-a meta-analysis. Med Sci Sports Exerc. 2014 Jun;46(6):1194-203. doi: 10.1249/MSS.0000000000000220. PMID 24576864
- [Background] Gualano B, Rawson ES, Candow DG, Chilibeck PD. Creatine supplementation in the aging population: effects on skeletal muscle, bone and brain. Amino Acids. 2016 Aug;48(8):1793-805. doi: 10.1007/s00726-016-2239-7. Epub 2016 Apr 23. PMID 27108136
- [Background] Pinto CL, Botelho PB, Carneiro JA, Mota JF. Impact of creatine supplementation in combination with resistance training on lean mass in the elderly. J Cachexia Sarcopenia Muscle. 2016 Sep;7(4):413-21. doi: 10.1002/jcsm.12094. Epub 2016 Jan 18. PMID 27239423
- [Background] Chilibeck PD, Kaviani M, Candow DG, Zello GA. Effect of creatine supplementation during resistance training on lean tissue mass and muscular strength in older adults: a meta-analysis. Open Access J Sports Med. 2017 Nov 2;8:213-226. doi: 10.2147/OAJSM.S123529. eCollection 2017. PMID 29138605
- [Background] Neves M Jr, Gualano B, Roschel H, Fuller R, Benatti FB, Pinto AL, Lima FR, Pereira RM, Lancha AH Jr, Bonfa E. Beneficial effect of creatine supplementation in knee osteoarthritis. Med Sci Sports Exerc. 2011 Aug;43(8):1538-43. doi: 10.1249/MSS.0b013e3182118592. PMID 21311365
- [Background] Bauer J, Biolo G, Cederholm T, Cesari M, Cruz-Jentoft AJ, Morley JE, Phillips S, Sieber C, Stehle P, Teta D, Visvanathan R, Volpi E, Boirie Y. Evidence-based recommendations for optimal dietary protein intake in older people: a position paper from the PROT-AGE Study Group. J Am Med Dir Assoc. 2013 Aug;14(8):542-59. doi: 10.1016/j.jamda.2013.05.021. Epub 2013 Jul 16. PMID 23867520
- [Background] Xu ZR, Tan ZJ, Zhang Q, Gui QF, Yang YM. The effectiveness of leucine on muscle protein synthesis, lean body mass and leg lean mass accretion in older people: a systematic review and meta-analysis. Br J Nutr. 2015 Jan 14;113(1):25-34. doi: 10.1017/S0007114514002475. Epub 2014 Sep 19. PMID 25234223
- [Background] Paddon-Jones D, Rasmussen BB. Dietary protein recommendations and the prevention of sarcopenia. Curr Opin Clin Nutr Metab Care. 2009 Jan;12(1):86-90. doi: 10.1097/MCO.0b013e32831cef8b. PMID 19057193
- [Background] Komar B, Schwingshackl L, Hoffmann G. Effects of leucine-rich protein supplements on anthropometric parameter and muscle strength in the elderly: a systematic review and meta-analysis. J Nutr Health Aging. 2015 Apr;19(4):437-46. doi: 10.1007/s12603-014-0559-4. PMID 25809808
- [Background] Wright AA, Cook CE, Baxter GD, Dockerty JD, Abbott JH. A comparison of 3 methodological approaches to defining major clinically important improvement of 4 performance measures in patients with hip osteoarthritis. J Orthop Sports Phys Ther. 2011 May;41(5):319-27. doi: 10.2519/jospt.2011.3515. Epub 2011 Feb 18. PMID 21335930
- [Background] Kreider RB, Kalman DS, Antonio J, Ziegenfuss TN, Wildman R, Collins R, Candow DG, Kleiner SM, Almada AL, Lopez HL. International Society of Sports Nutrition position stand: safety and efficacy of creatine supplementation in exercise, sport, and medicine. J Int Soc Sports Nutr. 2017 Jun 13;14:18. doi: 10.1186/s12970-017-0173-z. eCollection 2017. PMID 28615996